CLINICAL TRIAL: NCT00277303
Title: A Phase 2 Study of XL999 Administered Intravenously to Subjects With Metastatic Colorectal Cancer
Brief Title: Study of XL999 in Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to cardiac toxicities in the subjects
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W. Finn, PhD, President and CEO, Symphony Evolution, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL999-206
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Colorectal Cancer
Keywords: Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL999 — XL999 will be administered at 2.4 mg/kg as a 4-hour intravenous (IV) infusion. Subjects will receive XL999 infusions weekly for 8 weeks of treatment unless drug-related toxicity requires dosing delay. In the absence of progressive disease and unacceptable toxicity, subjects may receive XL999 treatment weekly for up to a year on this study. After 8 weeks, at the discretion of the investigator, one dose of four may be omitted for a subject's convenience.

SUMMARY:
This clinical study is being conducted at multiple sites to determine the activity, safety, and tolerability of XL999 when given weekly to patients with metastatic colorectal cancer (CRC). XL999 is a small molecule inhibitor of multiple kinases including VEGFR, PDGFR, FGFR, FLT-3, and Src, which are involved in tumor cell growth, formation of new blood vessels (angiogenesis), and metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with histologically confirmed metastatic colorectal cancer
* Measurable disease according to Response Criteria for Solid Tumors (RECIST)
* At least 1 prior therapeutic regimen (chemotherapy or biologic)
* ECOG performance status of 0 or 1
* Life expectancy ≥3 months
* Adequate organ and marrow function
* No other malignancies within 5 years
* Signed informed consent

Exclusion Criteria:

* Radiation to ≥25% of bone marrow within 30 days of XL999 treatment
* Treatment with systemic anticancer therapy within 30 days of XL999 treatment
* Subject has not recovered to ≤ grade 1 or to within 10% of baseline from adverse events due to other medications administered >30 days prior to study enrollment
* History of or known brain metastases, current spinal cord compression, or carcinomatous meningitis
* Uncontrolled and/or intercurrent illness
* Pregnant or breastfeeding females
* Known HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-12; Primary Completion 2006-08 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Response rate | Inclusion until disease progression
Safety and tolerability | Inclusion until 30 days post last treatment

SECONDARY OUTCOMES:
Progression-free survival | Inclusion until disease progression
Duration of response | Inclusion until disease progression
Overall survival | Inclusion until last Follow-up post last treatment or death
Pharmacokinetic (PK) and Pharmacodynamic (PD) parameters | Samples will be collected pre-dose and immediately at the end for subjects in the second stage of the study

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Bui, MD, Study Director — Exelixis
Locations (8):
- United States (8):
  - California Cancer Care, Inc., Greenbrae, California
  - Integrated Community Oncology Network; Division of Clinical Research, Jacksonville, Florida
  - Hematology Oncology Associated of the Treasure Coast, Port Saint Lucie, Florida
  - University of Chicago, Chicago, Illinois
  - Joliet Oncology-Hematology Associated, Ltd., Joliet, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Hematology Oncology Associates of Rockland, PC, New City, New York
  - Center for Oncology Research and Treatment, PA, Dallas, Texas